CLINICAL TRIAL: NCT00152503
Title: An Open Label, Exploratory, Dose-escalation, Multicenter Study Examining the Safety, Tolerability and Efficacy of Ucb 44212 (Seletracetam) Used at Doses of 10, 20, 40, and 80 mg b.i.d. (Total Daily Doses of 20 - 160 mg) Administration (Oral Capsules) in Adult Subjects (18 - 65 Years) With Refractory Epilepsy Suffering From Partial Onset Seizures Who Are Currently Receiving Levetiracetam (LEV) But Still Experiencing Seizures
Brief Title: Study With Subjects 18-65 Years Old With Partial Onset Seizures Who Are Currently Taking Levetiracetam
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma SA (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N01192
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Results first posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2022-10

CONDITIONS: Epilepsy, Partial
Keywords: Epilepsy; Partial Onset Seizures; Seletracetam; Levetiracetam
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy | interventions — Seletracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Seletracetam (Experimental): Escalating doses twice daily were to be administered.
  Interventions: Drug: Seletracetam (UCB44212)

INTERVENTIONS:
Drug: Seletracetam (UCB44212) — * Pharmaceutical form: oral capsules
  * Concentration: 2, 10 and 50 mg
  * Route of administration: oral administration

SUMMARY:
This trial will evaluate the efficacy and safety of UCB44212 as add-on therapy in subjects with focal epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Males/Females from 18 to 65 years of age (minimum body weight of 40 kg)
* Subjects with a confirmed diagnosis of epilepsy suffering from partial onset seizures whether or not secondarily generalized
* Subjects who have been treated for epilepsy for >= 6 months and are currently uncontrolled while being treated with 1-3 concomitant AED(s), inclusive of levetiracetam (LEV)
* Female subjects without childbearing potential or those who are using an acceptable contraceptive method

Exclusion Criteria:

* Seizures occurring in clusters. Status epilepticus within 6 months of Visit 1. History of non-epileptic seizures
* Subjects on vigabatrin
* Subjects on felbamate, unless treatment has been continuous for >2 years
* Ongoing psychiatric disease other than mild controlled disorders
* Subjects with clinically significant organ dysfunction
* Known allergic reaction or intolerance to pyrrolidine derivatives and/or excipients
* Pregnant or lactating women
* Use of benzodiazepines (for any indication) taken at a higher frequency than an average of once a week, unless counted as one of the concomitant Antiepileptic Drug (AEDs).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2005-08-31 (Actual); Primary Completion 2006-05-12 (Actual); Study Completion 2006-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — UCB (+1 844 599 2273)
Locations (17):
- United States (14):
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - St. Petersburg, Florida
  - Springfield, Illinois
  - Wichita, Kansas
  - Detroit, Michigan
  - Chesterfield, Missouri
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Dallas, Texas
  - Charlottesville, Virginia
  - Milwaukee, Wisconsin
- Canada (3):
  - Edmonton, Alberta
  - Calgary
  - Montreal

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in August 2005 and concluded in May 2006.
Pre-assignment Details: Participant Flow refers to the Intention-To-Treat Set. The study consisted of a 4-week Baseline Period, a 11-week Treatment Period (Up-/Down-Titration) and a 2-week Post-Treatment Period. Patients were up-titrated every two weeks until the maximum tolerated dose was reached. They were maintained at this dose until the end of the 8-week Up-Titration Period and continue that dose until the Down-Titration Visit scheduled for that dose level. Patients were to be down-titrated over a 3-week Period.
Groups:
- Seletracetam: Escalating doses of 10, 20, 40 and 80 mg b.i.d. (twice daily) (total daily doses of 20 - 160 mg) were to be administered orally as capsules.
Period: Overall Study
Arm/Group | Seletracetam
Started | 59
Completed | 55
Not Completed | 4
Not completed — Adverse Event | 4

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Intention-to-Treat (ITT) population.
Arm/Group | Seletracetam
Number analyzed (Participants) | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 59
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.34 (10.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 28

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Seizure Frequency Per Week for Partial Onset Seizures (Type I) by Visit and Overall by Period
Description: Calculated as (7-day seizure frequency during the Treatment Period) - (7-day seizure frequency during the Baseline Period (Week 1 to Week 4)), divided by the 7-day seizure frequency during the Baseline Period with this quantity multiplied by 100. A negative value in percent change from Baseline indicates a decrease in partial onset seizure frequency from Baseline.
  The Treatment Period consists of an 8-week Up-Titration Period (Visit 3/Week 5 to Visit 7/Week 12) and a 3-week Down-Titration Period (Visit 7/Week 13 to Visit 10/Week 15). Visit x includes the period from the beginning of Visit x-1 up to but not including Visit x.
Time Frame: During the Treatment Period (Week 5 to Week 15), compared to Baseline Period (Week 1 to Week 4)
Population: 59 subjects were included in the ITT-set, who took at least one dose of trial medication. Only subjects with available data for the respective visit/ period are included in the analysis. Number of subjects analyzed is given separately for each visit/ period.
Measure: Median (Inter-Quartile Range); unit: percentage of change
Arm/Group | Seletracetam
Number analyzed (Participants) | 59
percentage of change
  Visit 4 (Week 5 and 6): number analyzed (Participants) | 56
  Visit 4 (Week 5 and 6) | -26.07 [-49.29 to -5.88]
  Visit 5 (Week 7 and 8): number analyzed (Participants) | 56
  Visit 5 (Week 7 and 8) | -32.05 [-52.60 to -8.46]
  Visit 6 (Week 9 and 10): number analyzed (Participants) | 55
  Visit 6 (Week 9 and 10) | -42.22 [-66.67 to -25.00]
  Visit 7 (Week 11 and 12): number analyzed (Participants) | 56
  Visit 7 (Week 11 and 12) | -31.67 [-79.00 to 9.02]
  Up-titration (Weeks 5 to 12): number analyzed (Participants) | 56
  Up-titration (Weeks 5 to 12) | -34.01 [-50.69 to -13.27]
  Visit 8 (Week 13): number analyzed (Participants) | 55
  Visit 8 (Week 13) | -44.44 [-74.60 to -10.00]
  Visit 9 (Week 14): number analyzed (Participants) | 55
  Visit 9 (Week 14) | -22.22 [-55.56 to 12.50]
  Visit 10 (Week 15): number analyzed (Participants) | 54
  Visit 10 (Week 15) | -33.85 [-61.79 to 35.00]
  Down-titration (Weeks 13 to 15): number analyzed (Participants) | 55
  Down-titration (Weeks 13 to 15) | -29.29 [-51.05 to 6.06]
  On Treatment (Weeks 5 to 15): number analyzed (Participants) | 56
  On Treatment (Weeks 5 to 15) | -33.09 [-47.38 to -13.20]

2. Secondary Outcome: Percent Change From Baseline in Seizure Frequency Per Week for All Seizure Types (Types I + II + III) by Visit and Overall by Period
Description: Calculated as (7-day seizure frequency during the Treatment Period) - (7-day seizure frequency during the Baseline Period (Week 1 to Week 4)), divided by the 7-day seizure frequency during the Baseline Period with this quantity multiplied by 100. A negative value in percent change from Baseline indicates a decrease in seizure frequency from Baseline.
  The Treatment Period consists of an 8-week Up-Titration Period (Visit 3/Week 5 to Visit 7/Week 12) and a 3-week Down-Titration Period (Visit 7/Week 13 to Visit 10/Week 15). Visit x includes the period from the beginning of Visit x-1 up to but not including Visit x.
Time Frame: During the Treatment Period (Week 5 to Week 15), compared to Baseline Period (Week 1 to Week 4)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of change
Arm/Group | Seletracetam
Number analyzed (Participants) | 59
percentage of change
  Visit 4 (Week 5 and 6): number analyzed (Participants) | 56
  Visit 4 (Week 5 and 6) | -26.07 [-49.29 to -5.88]
  Visit 5 (Week 7 and 8): number analyzed (Participants) | 56
  Visit 5 (Week 7 and 8) | -32.05 [-52.60 to -8.46]
  Visit 6 (Week 9 and 10): number analyzed (Participants) | 55
  Visit 6 (Week 9 and 10) | -42.22 [-66.67 to -25.00]
  Visit 7 (Week 11 and 12): number analyzed (Participants) | 56
  Visit 7 (Week 11 and 12) | -31.67 [-79.00 to 9.02]
  Up-titration (Weeks 5 to 12): number analyzed (Participants) | 56
  Up-titration (Weeks 5 to 12) | -34.01 [-50.69 to -13.27]
  Visit 8 (Week 13): number analyzed (Participants) | 55
  Visit 8 (Week 13) | -44.44 [-74.60 to -10.00]
  Visit 9 (Week 14): number analyzed (Participants) | 55
  Visit 9 (Week 14) | -22.22 [-55.56 to 12.50]
  Visit 10 (Week 15): number analyzed (Participants) | 54
  Visit 10 (Week 15) | -33.85 [-61.79 to 35.00]
  Down-Titration (Weeks 13 to 15): number analyzed (Participants) | 55
  Down-Titration (Weeks 13 to 15) | -29.29 [-51.05 to 6.06]
  On Treatment (Weeks 5 to 15): number analyzed (Participants) | 55
  On Treatment (Weeks 5 to 15) | -33.09 [-47.38 to -13.20]

3. Secondary Outcome: Change From Baseline in Seizure Frequency Per Week for Partial Onset Seizures (Type I) by Visit and Overall by Period
Description: as for outcome 1
Time Frame: During the Treatment Period (Week 5 to Week 15), compared to Baseline Period (Week 1 to Week 4)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: seizures per week
Arm/Group | Seletracetam
Number analyzed (Participants) | 59
seizures per week
  Visit 4 (Week 5 and 6): number analyzed (Participants) | 56
  Visit 4 (Week 5 and 6) | -0.85 [-2.92 to -0.17]
  Visit 5 (Week 7 and 8): number analyzed (Participants) | 56
  Visit 5 (Week 7 and 8) | -1.25 [-3.22 to -0.39]
  Visit 6 (Week 9 and 10): number analyzed (Participants) | 55
  Visit 6 (Week 9 and 10) | -1.83 [-3.13 to -0.68]
  Visit 7 (Week 11 and 12): number analyzed (Participants) | 56
  Visit 7 (Week 11 and 12) | -1.31 [-3.13 to 0.27]
  Up-titration (Weeks 5 to 12): number analyzed (Participants) | 56
  Up-titration (Weeks 5 to 12) | -1.36 [-2.77 to -0.56]
  Visit 8 (Week 13): number analyzed (Participants) | 55
  Visit 8 (Week 13) | -1.68 [-3.63 to -0.31]
  Visit 9 (Week 14): number analyzed (Participants) | 55
  Visit 9 (Week 14) | -1.00 [-2.63 to 0.48]
  Visit 10 (Week 15): number analyzed (Participants) | 54
  Visit 10 (Week 15) | -1.14 [-3.11 to 1.38]
  Down-Titration (Weeks 13 to 15): number analyzed (Participants) | 55
  Down-Titration (Weeks 13 to 15) | -1.09 [-2.30 to 0.25]
  On Treatment (Weeks 5 to 15): number analyzed (Participants) | 56
  On Treatment (Weeks 5 to 15) | -1.13 [-2.62 to -0.49]

4. Secondary Outcome: Change From Baseline in Seizure Frequency Per Week for All Seizure Types (Types I + II + III) by Visit and Overall by Period
Description: as for outcome 2
Time Frame: During the Treatment Period (Week 5 to Week 15), compared to Baseline Period (Week 1 to Week 4)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: seizures per week
Arm/Group | Seletracetam
Number analyzed (Participants) | 59
seizures per week
  Visit 4 (Week 5 and 6): number analyzed (Participants) | 56
  Visit 4 (Week 5 and 6) | -0.85 [-2.92 to -0.17]
  Visit 5 (Week 7 and 8): number analyzed (Participants) | 56
  Visit 5 (Week 7 and 8) | -1.25 [-3.22 to -0.39]
  Visit 6 (Week 9 and 10): number analyzed (Participants) | 55
  Visit 6 (Week 9 and 10) | -1.83 [-3.13 to -0.68]
  Visit 7 (Week 11 and 12): number analyzed (Participants) | 56
  Visit 7 (Week 11 and 12) | -1.31 [-3.13 to 0.27]
  Up-titration (Weeks 5 to 12): number analyzed (Participants) | 56
  Up-titration (Weeks 5 to 12) | -1.36 [-2.77 to -0.56]
  Visit 8 (Week 13): number analyzed (Participants) | 55
  Visit 8 (Week 13) | -1.68 [-3.63 to -0.31]
  Visit 9 (Week 14): number analyzed (Participants) | 55
  Visit 9 (Week 14) | -1.00 [-2.63 to 0.48]
  Visit 10 (Week 15): number analyzed (Participants) | 54
  Visit 10 (Week 15) | -1.14 [-3.11 to 1.38]
  Down-Titration (Weeks 13 to 15): number analyzed (Participants) | 55
  Down-Titration (Weeks 13 to 15) | -1.09 [-2.30 to 0.25]
  On Treatment (Weeks 5 to 15): number analyzed (Participants) | 55
  On Treatment (Weeks 5 to 15) | -1.13 [-2.62 to -0.49]

5. Secondary Outcome: Seizure Frequency Per Week (Type I) by Visit Over the Treatment Period and Overall by Period
Description: Calculated as 7-day partial onset seizure (type I) frequency; The Treatment Period consists of an 8-week Up-Titration Period (Visit 3/Week 5 to Visit 7/Week 12) and a 3-week Down-Titration Period (Visit 7/Week 13 to Visit 10/Week 15). Visit x includes the period from the beginning of Visit x-1 up to but not including Visit x.
Time Frame: During the Treatment Period (Week 5 to Week 15)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: seizure frequency per week
Arm/Group | Seletracetam
Number analyzed (Participants) | 59
seizure frequency per week
  Baseline (Week 1 to Week 4) | 3.63 [2.42 to 7.50]
  Visit 4 (Week 5 and 6): number analyzed (Participants) | 56
  Visit 4 (Week 5 and 6) | 3.25 [1.57 to 5.96]
  Visit 5 (Week 7 and 8): number analyzed (Participants) | 56
  Visit 5 (Week 7 and 8) | 2.90 [1.50 to 5.19]
  Visit 6 (Week 9 and 10): number analyzed (Participants) | 55
  Visit 6 (Week 9 and 10) | 2.15 [1.08 to 8.40]
  Visit 7 (Week 11 and 12): number analyzed (Participants) | 56
  Visit 7 (Week 11 and 12) | 2.27 [0.74 to 5.67]
  Up-titration (Weeks 5 to 12): number analyzed (Participants) | 56
  Up-titration (Weeks 5 to 12) | 2.71 [1.56 to 6.40]
  Visit 8 (Week 13): number analyzed (Participants) | 55
  Visit 8 (Week 13) | 2.63 [1.00 to 5.00]
  Visit 9 (Week 14): number analyzed (Participants) | 55
  Visit 9 (Week 14) | 3.00 [1.17 to 9.00]
  Visit 10 (Week 15): number analyzed (Participants) | 54
  Visit 10 (Week 15) | 3.50 [1.40 to 8.75]
  Down-Titration (Weeks 13 to 15): number analyzed (Participants) | 55
  Down-Titration (Weeks 13 to 15) | 3.18 [1.59 to 7.00]
  On Treatment (Weeks 5 to 15): number analyzed (Participants) | 56
  On Treatment (Weeks 5 to 15) | 3.02 [1.67 to 6.20]

6. Secondary Outcome: Seizure Frequency Per Week (Type I+II+III) by Visit Over the Treatment Period and Overall by Period
Description: Calculated as 7-day seizure frequency for all seizure types (type I+II+III). The Treatment Period consists of an 8-week Up-Titration Period (Visit 3/Week 5 to Visit 7/Week 12) and a 3-week Down-Titration Period (Visit 7/Week 13 to Visit 10/Week 15). Visit x includes the period from the beginning of Visit x-1 up to but not including Visit x.
Time Frame: During the Treatment Period (Week 5 to Week 15)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: seizure frequency per week
Arm/Group | Seletracetam
Number analyzed (Participants) | 59
seizure frequency per week
  Baseline (Week 1 to Week 4) | 3.63 [2.42 to 7.50]
  Visit 4 (Week 5 and 6): number analyzed (Participants) | 56
  Visit 4 (Week 5 and 6) | 3.25 [1.57 to 5.96]
  Visit 5 (Week 7 and 8): number analyzed (Participants) | 56
  Visit 5 (Week 7 and 8) | 2.90 [1.50 to 5.19]
  Visit 6 (Week 9 and 10): number analyzed (Participants) | 55
  Visit 6 (Week 9 and 10) | 2.15 [1.08 to 8.40]
  Visit 7 (Week 11 and 12): number analyzed (Participants) | 56
  Visit 7 (Week 11 and 12) | 2.27 [0.74 to 5.67]
  Up-titration (Weeks 5 to 12): number analyzed (Participants) | 56
  Up-titration (Weeks 5 to 12) | 2.71 [1.56 to 6.40]
  Visit 8 (Week 13): number analyzed (Participants) | 55
  Visit 8 (Week 13) | 2.63 [1.00 to 5.00]
  Visit 9 (Week 14): number analyzed (Participants) | 55
  Visit 9 (Week 14) | 3.00 [1.17 to 9.00]
  Visit 10 (Week 15): number analyzed (Participants) | 54
  Visit 10 (Week 15) | 3.50 [1.40 to 8.75]
  On Treatment (Weeks 5 to 15): number analyzed (Participants) | 56
  On Treatment (Weeks 5 to 15) | 3.02 [1.67 to 6.20]
  Down-Titration (Weeks 13 to 15): number analyzed (Participants) | 55
  Down-Titration (Weeks 13 to 15) | 3.18 [1.59 to 7.00]

7. Secondary Outcome: Percentage of Responder Subjects in Partial Onset Seizures (Type I) Over the Up-titration Period
Description: A responder was defined as a subject with a >= 50% reduction in seizure frequency per week from the Baseline Period (Week 1 to Week 4) to the end of the Up-Titration Period.
Time Frame: During the Up-Titration Period (Week 5 to Week 12), compared to Baseline Period (Week 1 to Week 4)
Population: 59 subjects were included in the ITT-set, who took at least one dose of trial medication. Only subjects with available post-baseline seizure data are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Seletracetam
Number analyzed (Participants) | 56
percentage of participants | 28.6

8. Secondary Outcome: Categorized Percentage Response to Treatment in Partial Onset Seizures (Type I) Over the Up-titration Period
Description: Response to treatment in partial onset seizures (type I) over the up-titration period were analyzed by the percentage change from baseline (Week 1 to Week 4) in partial seizure frequency per week over the up-titration period, grouped in 4 categories: <-25%, -25% to <25%, 25% to <75%, and 75% to 100%.
Time Frame: During the Up-Titration Period (Week 5 to Week 12), compared to Baseline Period (Week 1 to Week 4)
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Seletracetam
Number analyzed (Participants) | 56
percentage of participants
  < -25% | 12.5
  -25% to < 25% | 25.0
  25% to < 75% | 57.1
  75% to <100% | 5.4

9. Secondary Outcome: Percent Change From Baseline in Seizure-free Days Per Week Over the Up-titration Period
Description: A day was considered seizure-free, if no seizure was reported during 24 hours. A positive value indicates improvement from Baseline (Week 1 to Week 4).
Time Frame: During the Up-Titration Period (Week 5 to Week 12), compared to Baseline Period (Week 1 to Week 4)
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: percentage of change
Arm/Group | Seletracetam
Number analyzed (Participants) | 52
percentage of change | 11.45 [1.45 to 28.99]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Baseline to Follow-Up visit (up to Week 17).
Description: Adverse Events refer to the Intention-To-Treat (ITT) population.
Arm/Group | Seletracetam
All-Cause Mortality (participants affected / at risk) | 0/59
Serious Adverse Events (participants affected / at risk) | 2/59
Other Adverse Events (participants affected / at risk) | 44/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Seletracetam (N=59)
Angina unstable (Cardiac disorders) | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Convulsion (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Seletracetam (N=59)
Abdominal pain upper (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 12
Vomiting (Gastrointestinal disorders) | 6
Fatigue (General disorders) | 8
Irritability (General disorders) | 3
Bronchitis (Infections and infestations) | 3
Herpes simplex (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 7
Upper respiratory tract infection (Infections and infestations) | 6
Decreased appetite (Metabolism and nutrition disorders) | 3
Convulsion (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 13
Headache (Nervous system disorders) | 9
Nystagmus (Nervous system disorders) | 4
Somnolence (Nervous system disorders) | 8
Tremor (Nervous system disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days